CLINICAL TRIAL: NCT02096705
Title: A 24-week Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 3 Trial to Evaluate Efficacy and Safety of Dapagliflozin Added to Therapy of Asian Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Insulin
Brief Title: Phase III Insulin Add-On Asia Regional Program - ST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB102-137
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: Dapagliflozin (Experimental): Dapagliflozin 10 mg oral Tablet once daily for 24 weeks + Background Insulin
  Interventions: Drug: Dapagliflozin
- Group 2: Dapagliflozin Placebo (Placebo Comparator): Dapagliflozin Placebo 0 mg oral Tablet once daily for 24 weeks + Background Insulin
  Interventions: Drug: Dapagliflozin Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Tablet
  Other Names: BMS-512148
  Arms: Group 1: Dapagliflozin
Drug: Dapagliflozin Placebo — Tablet
  Arms: Group 2: Dapagliflozin Placebo

SUMMARY:
The purpose is to determine if after 24 weeks of oral daily administration, there will be a greater mean reduction from baseline in glycosylated hemoglobin (HbA1c) achieved with Dapagliflozin 10 mg plus insulin compared to placebo plus insulin in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have type 2 diabetes with inadequate glycemic control, defined as HbA1c ≥ 7.5% and ≤ 11.0% obtained at screening visit
* Subjects must be taking a stable mean dose of ≥ 20 IU injectable insulin daily for at least 8 weeks prior to enrollment

Inclusion criteria for randomization:

HbA1c ≥ 7.5 and ≤ 10.5% at Day -14

Exclusion Criteria:

* Treatment with more than two oral antidiabetic (OAD) agents within 6 weeks of Enrollment
* History of diabetic ketoacidosis of hyperosmolar nonketotic coma
* Clinically diagnosed Type 1 diabetes mellitus
* Congestive heart failure defined as New York Heart Association (NYHA) stage III and IV
* Severe uncontrolled hypertension defined as systolic blood pressure (SBP) ≥ 180 mmHg and/or diastolic blood pressure (DBP) ≥ 110 mmHg
* History of unstable or rapidly progressing renal disease
* History of severe hepatobiliary disease
* Mallingancy within 5 years of the screening/enrollment visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2016-01-28 (Actual); Study Completion 2016-01-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- China (14):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Haerbin, Heilongjiang
  - Local Institution, Changsha, Hunan
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Suzhou, Jiangsu
  - Local Institution, Wuxi, Jiangsu
  - Local Institution, Changchun, Jilin
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Xi’an, Shanxi
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Chongqing, Sichuan
  - Local Institution, Beijing
  - Local Institution, Tianjin
- Local Institution, Singapore, Singapore
- South Korea (4):
  - Local Institution, Busan
  - Local Institution, Daegu
  - Local Institution, Daejeon
  - Local Institution, Seoul

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 477 participants were enrolled; 313 entered lead-in period; 272 participants were randomized to a treatment group. Of the 205 participants not randomized to a treatment group: 190 No longer met study criteria, 11 withdrew consent, 2 were lost to follow-up, and 2 were removed for administrative reasons.
Groups:
- Placebo: Dapagliflozin Placebo 0 mg oral Tablet once daily for 24 weeks + Background Insulin
- Dapagliflozin: Dapagliflozin 10 mg oral Tablet once daily for 24 weeks + Background Insulin
Period: Treatment
Arm/Group | Placebo | Dapagliflozin
Started | 133 | 139
Completed | 124 | 134
Not Completed | 9 | 5
Not completed — Adverse Event | 6 | 3
Not completed — Subject request to discontinue treatment | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 1 | 1
Period: Follow-up
Arm/Group | Placebo | Dapagliflozin
Started | 129 (5 participants in this arm did not complete the treatment period and rejoined for follow-up) | 139 (5 participants in this arm did not complete the treatment period and rejoined for follow-up)
Completed | 125 | 135
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 2 | 2
Not completed — Subjects not reporting status | 1 | 2

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dapagliflozin | Total
Number analyzed (Participants) | 133 | 139 | 272
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 117 | 214
  >=65 years | 36 | 22 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (8.91) | 56.5 (8.39) | 57.5 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 73 | 142
  Male | 64 | 66 | 130

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change in HbA1c From Baseline to Week 24
Description: The adjusted mean change in the percentage of Hemoglobin A1c (HbA1c) from baseline to Week 24 was reported for each arm.
Time Frame: Baseline (Day 1) and 24 weeks
Population: All randomized participants with non-missing baseline and at least one post-baseline value
Measure: Mean (Standard Error); unit: percentage of hemoglobin
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 129 | 137
percentage of hemoglobin | 0.03 (0.0707) | -0.87 (0.0666)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin; Test type: Superiority or Other; p < 0.0001, Longitudinal repeated measure analysis — P-value for Dapagliflozin vs. placebo; Mean Difference (Final Values) = -0.90, 95% CI 2-sided [-1.09 to -0.71], Standard Error of Mean 0.0968 — Difference of Dapagliflozin from placebo

2. Secondary Outcome: Adjusted Mean Change in Fasting Plasma Glucose (FPG) From Baseline to Week 24
Description: The adjusted mean change from baseline to 24 weeks in Fasting Plasma Glucose (FPG) was reported for each arm in milligrams per deciliter (mg/dL).
Time Frame: Baseline (Day 1) and 24 weeks
Population: All randomized participants with non-missing baseline and at least one post-baseline value
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 133 | 138
mg/dL | 0.07 (3.3803) | -30.62 (3.1314)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin; Test type: Superiority or Other; p < 0.0001, Longitudinal repeated measure analysis; P-value for Dapagliflozin vs. placebo; Mean Difference (Final Values) = -30.69, 95% CI 2-sided [-39.76 to -21.61], Standard Error of Mean 4.6050 — Difference of Dapagliflozin from placebo

3. Secondary Outcome: Adjusted Mean Change in Body Weight From Baseline to Week 24
Description: Adjusted mean change in body weight from baseline to week 24 was reported for each arm in kilograms (kg).
Time Frame: Baseline (Day 1) and 24 weeks
Population: All randomized participants with non-missing baseline and at least one post-baseline value
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 133 | 138
kilograms | 0.37 (0.2224) | -1.00 (0.2103)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin; Test type: Superiority or Other; p < 0.0001, Longitudinal repeated measure analysis — P-value for Dapagliflozin vs. placebo; Mean Difference (Final Values) = -1.38, 95% CI 2-sided [-1.98 to -0.77], Standard Error of Mean 0.3057 — Difference of Dapagliflozin from placebo

4. Secondary Outcome: Adjusted Mean Change in Absolute Calculated Mean Total Daily Dose of Insulin (TDDI) From Baseline to Week 24
Description: The adjusted mean change in absolute calculated mean Total Daily Dose of Insulin (TDDI) from baseline to week 24 was reported for each arm in International Units (IU).
Time Frame: Baseline (Day 1) and 24 weeks
Population: All randomized participants with non-missing baseline and at least one post-baseline value
Measure: Mean (Standard Error); unit: International Units (IU)
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 133 | 139
International Units (IU) | 0.74 (0.3723) | -0.70 (0.3592)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin; Test type: Superiority or Other; p = 0.0059, Longitudinal repeated measure analysis — P-value for Dapagliflozin vs. placebo; Mean Difference (Final Values) = -1.43, 95% CI 2-sided [-2.45 to -0.42], Standard Error of Mean 0.5171 — Difference of Dapagliflozin from placebo

ADVERSE EVENTS:
Time Frame: 24 week treatment period + 30 days
Description: Includes serious adverse events with onset on or after the first date/time of double-blind treatment and on or prior to the last day of double blind treatment plus 30 days. Includes non-serious adverse events with onset on or after the first date/time of double-blind treatment and on or prior to the last day of double blind treatment plus 4 days.
Arm/Group | Dapagliflozin | Placebo
Serious Adverse Events (participants affected / at risk) | 8/139 | 18/133
Other Adverse Events (participants affected / at risk) | 61/139 | 61/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=139) | Placebo (N=133)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL BRIDGING (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 0 (0) | 1 (1)
UVEITIS (Eye disorders) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 1 (1) | 0 (0)
NEUROSYPHILIS (Infections and infestations) | 0 (0) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ARACHNOID CYST (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
DIABETIC NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
VIITH NERVE PARALYSIS (Nervous system disorders) | 0 (0) | 1 (1)
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
CALCULUS URETERIC (Renal and urinary disorders) | 1 (1) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=139) | Placebo (N=133)
NASOPHARYNGITIS (Infections and infestations) | 5 (6) | 7 (8)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (8) | 9 (12)
URINARY TRACT INFECTION (Infections and infestations) | 5 (5) | 7 (7)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 9 (9) | 12 (13)
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 31 (36) | 31 (31)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 12 (13) | 12 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.